CLINICAL TRIAL: NCT04582708
Title: Use of NERv's Inline Device for the Continuous Monitoring of pH and Conductivity as an Early Diagnostic Method for Postoperative Complications
Brief Title: Use of NERv's Inline Device as an Early Diagnostic Method for Postoperative Complications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FluidAI Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLS0006
Record Dates: First submitted 2020-09-30; First posted 2020-10-09 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Anastomotic Leak; Fistula; Postoperative Leak; Postoperative Pancreatic Fistula; POPF
MeSH Terms: conditions — Anastomotic Leak; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with NERv's Inline Device Attached (Experimental): This arm contains subjects which will have NERv's Inline Device attached to their peritoneal drain after abdominal surgery.
  Interventions: Device: NERv's Inline Device

INTERVENTIONS:
Device: NERv's Inline Device — NERv's Inline Device is comprised of multiple sensors. It attaches in line to existing catheters or peritoneal drains that are currently approved for medical use. This allows the device to measure the pH and electrical conductivity of effluent fluids that are drained through peritoneal drains.

SUMMARY:
NERv's traditional feasibility clinical trial is a multi-center, pre-market, single-arm, and non-randomized trial. This study will involve the retrospective analysis of prospectively collected data. The trial is intended to establish the safety of NERv's Inline Device and collect preliminary data to illustrate the change in pH and electrical conductivity during normal postoperative recovery and in the event of a complication.

The purpose of NERv's feasibility study is to establish a clinical model that shows the progressive change in pH and electrical conductivity during a normal post-operative recovery and in the event of an anastomotic leak in colorectal, hepatobiliary (HPB), trauma, and general surgery patients. Upon analyzing data collected from NERv's Inline Device, a clinical model of change in pH and conductivity over time will be created. The clinical model can be used in future stages to determine if a complication is developing. For instance, boundaries (reading thresholds) can be established to detect a complication when readings exceed such boundaries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years - male or female
* Subject understands and has voluntarily signed and dated Informed Consent Form (ICF)
* Subjects must be willing to comply with trial requirements
* Subject has a peritoneal drain, such as Jackson Pratt drain attached post abdominal surgery

Exclusion Criteria:

* Plans that the subject will be discharged in less than 8 hours post-surgery
* Involvement in the planning and conduct of the clinical investigation
* Subject is participating in another investigational drug or device study which may interfere with the endpoints of this study
* NERv's Inline Device does not attach to drain used on the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Change in pH of Peritoneal Fluid | A clinical model of change in pH over time will be established once the study is completed (up to 18 months)
  NERv's Inline Device will be collecting continuous pH measurements of effluent fluid in abdominal surgery patients during normal recovery and in the event of a complication
Change in Electrical Conductivity of Peritoneal Fluid | A clinical model of change in electrical conductivity over time will be established once the study is completed (up to 18 months)
  NERv's Inline Device will be collecting continuous electrical conductivity measurements of effluent fluid in abdominal surgery patients during normal recovery and in the event of a complication
Number of Subjects with Device Related Adverse Events | The total number of device related adverse events will be established once the study is completed (up to 18 months)
  An adverse event assessment will be performed in accordance to ISO 14155 standards to determine the number of device related adverse events

SECONDARY OUTCOMES:
Investigator Feedback on Device's Ease of Use | Ease of use and impact on workflow will be established once the study is completed (up to 18 months)
  Ease of use and Impact on workflow will be evaluated by collecting responses to a questionnaire that will be filled out by the study team. The study team will evaluate the device's attachment, removal, setup, calibration, and their overall experience with the user interface on NERv's Mobile Application. The study team will be asked to rate their experience on a scale of 1-5, with 1 being very unsatisfied and 5 being very satisfied.
Subject Feedback on Device's Comfort level | Comfort level will be established once the study is completed (up to 18 months)
  Comfort level will be evaluated by collecting responses to a questionnaire that will be filled out by the subject. The subject will evaluate the device's weight, size, design, and their ability to sleep comfortably with the device attached. The subject will be asked to rate their experience on a scale of 1-5, with 1 being very unsatisfied and 5 being very satisfied.
Estimate the economic benefit of the early detection of anastomotic leaks by contrasting the time of detection using NERv's Inline Device and Standard of Care | The economic benefit of using NERv's Inline Device will be established once the study is completed (up to 18 months)
  Retrospective data analysis will be performed to estimate the economic benefit of early detection of anastomotic leaks in patients undergoing gastrointestinal procedures by comparing the time of detection using NERv's Inline device and the time of detection using standard of care

CONTACTS AND LOCATIONS:
Locations (7):
- Cleveland Clinic, Cleveland, Ohio, United States
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Juravinski Hospital- Hamilton Health Sciences, Hamilton, Ontrario
- King Saud University Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No